CLINICAL TRIAL: NCT01452958
Title: Endotoxin & Cytokines. Do Protein Loss and Metabolic Effects Depend on CNS Activation of Stress Hormones or on Local Mechanisms in Muscle and Fat?
Brief Title: Endotoxin & Cytokines. Do Protein Loss and Metabolic Effects Depend on Central Nervous System (CNS) Activation of Stress Hormones or on Local Mechanisms in Muscle and Fat?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aarhus University Hospital (Other)
Collaborators: University of Aarhus (Other); Lundbeck Foundation (Other)
Responsible Party: Principal Investigator, Ermina Bosnjak, Medical Doctor, PhD student, Aarhus University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: 2010/0604
Record Dates: First submitted 2011-09-22; First posted 2011-10-17 (Estimated); Last update posted 2013-01-30 (Estimated); Status verified 2013-01

CONDITIONS: Inflammation; Glucose Metabolism Disorders
Keywords: Endotoxin; LPS; TNF-α; insulin resistance; metabolism
MeSH Terms: conditions — Inflammation; Glucose Metabolism Disorders; Insulin Resistance | interventions — Tumor Necrosis Factor-alpha; Endotoxins

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TNF-α (Experimental): Beromun, Boehringer-Ingelheim, Germany
  Interventions: Biological: TNF-alpha
- Endotoxin (Experimental)
  Interventions: Biological: Endotoxin

INTERVENTIONS:
Biological: TNF-alpha — Study protocol 1: 6 ng/kg/h intraarterial Study protocol 2: 18 ng/kg/h intravenous
  Other Names: Beromun, Boehringer-Ingelheim, Germany
  Arms: TNF-α
Biological: Endotoxin — Study protocol 2:0,075 ng/kg/h intravenous
  Other Names: E. coli endotoxin, US standard
  Arms: Endotoxin

SUMMARY:
Main objective :

The purpose of this study is to prove that the effects of bacterial endotoxin and cytokine TNF-α, on protein loss, fatty acid release, and glucose metabolism depend on two mechanisms:

1. Direct local effects in muscle tissue.
2. Activation of the hypothalamo-pituitary axis and a stress-hormone response

Study protocols:

1. Acute metabolic effects of TNF-α(Beromun, Boehringer-Ingelheim Germany) vs placebo perfused into the femoral artery of the leg in 8 healthy subjects.
2. Acute metabolic effects of

   * placebo(saline)
   * endotoxin(US standard reference E.Coli, endotoxin)
   * TNF-α(Beromun, Boehringer-Ingelheim Germany) given systemically
   * in 8 patients with hypopituitarism(to block stress hormone release) and in 8 healthy subjects all studied thrice.

DETAILED DESCRIPTION:
PURPOSE:

Knowledge about the effects of bacterial endotoxin and cytokines (and inflammation in general) in humans on protein, glucose and lipid metabolism and intracellular signalling in muscle and fat is sporadic and it is uncertain whether endotoxin and cytokines act directly in fat and muscle tissue or indirectly via central nervous system (CNS) mediated stress hormone release.

The investigators hypothesize that the metabolic effects of endotoxin and cytokine TNF-α, including protein loss, fatty acid release and decreased glucose uptake depend on two mechanisms:

1. Direct local effects in muscle tissue (Study protocol 1)
2. Activation of the hypothalamo-pituitary axis and generalized stress hormone response (Study protocol 2)

METHODOLOGY:

Study protocol 1:

Acute metabolic effects of TNF-α (Beromun, Boehringer-Ingelheim, Germany) versus placebo perfused into the femoral artery of the leg in 8 healthy subjects, studied once. Femoral vein sampling allows assessment of local metabolic events in the leg. The vessels were cannulated using the Seldinger technique. Each study comprises a 3 hour basal period and a 3 hour Hyperinsulinemic-Euglycemic Clamp. Muscle biopsies were obtained simultaneously from both lateral vastus muscles.

Study protocol 2:

Acute metabolic effects of (i)placebo (saline), (ii)endotoxin (US standard reference E.Coli, endotoxin) and (iii)TNF-α (Beromun, Boehringer-Ingelheim, Germany) given systemically intravenously (i.v.) in 8 patients with hypopituitarism (to block stress hormone release) and in 8 healthy subjects all studied thrice. Every study comprises a 4 hour basal period and a 2 hour Hyperinsulinemic-Euglycemic Clamp. Muscle and fat biopsies were obtained.

Study protocol 1 and Study protocol 2:

Assays: Mass spectrometry (15N-phenylalanine, 13C-urea), 3H-glucose, 3H-palmitate quantification, hormone and metabolite analysis, cytokine assays, intracellular signaling.

ELIGIBILITY:
Inclusion Criteria 1. group:

* Male
* 19 < BMI < 28
* 18 ≤ Age ≤ 50
* Healthy

Inclusion Criteria 2. group:

* Male
* 20 < BMI < 30
* Age > 25
* Healthy

Exclusion Criteria:

* Diseases
* Allergy

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2010-06; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Acute metabolic effects of endotoxin and cytokine TNF-α (Study 2) | 2 hours
  During a basal period.
  Acute metabolic effects: Glucose metabolism was quantified with raw arterio-venous differences and 3H3-Glucose tracer. Lactate was quantified with raw arterio-venous differences. Lipid metabolism was quantified with [9,10-3H]-Palmitate tracer and amino acid metabolism with 15N-Phenylalanine tracer and 13C-Urea tracer.
Acute metabolic effects of endotoxin and cytokine TNF-α (Study 2) | 4 hours
  During a hyperinsulinaemic euglycaemic clamp.
  Acute metabolic effects: Glucose metabolism was quantified with raw arterio-venous differences and 3H3-Glucose tracer. Lactate was quantified with raw arterio-venous differences. Lipid metabolism was quantified with [9,10-3H]-Palmitate tracer and amino acid metabolism with 15N-Phenylalanine tracer and 13C-Urea tracer.
Acute metabolic effects of cytokine TNF-α (Study 1) | 3 hours
  During a basal period.
  Acute metabolic effects: Glucose and lactate were quantified with raw arterio-venous differences; lipid metabolism was quantified with [9,10-3H]-palmitate and amino acid metabolism with 15N-phenylalanine.
Acute metabolic effects of cytokine TNF-α (Study 1) | 3 hours
  During a hyperinsulinaemic euglycaemic clamp.
  Acute metabolic effects: Glucose and lactate were quantified with raw arterio-venous differences; lipid metabolism was quantified with [9,10-3H]-palmitate and amino acid metabolism with 15N-phenylalanine.

SECONDARY OUTCOMES:
Intracellular insulin signaling, growth hormone signalling and inflammatory signalling pathways. | 120 min.
  Musle and fat biopsies during a basal period (120 min. from the beginning of a basal period)
Intracellular insulin signaling, growth hormone signalling and inflammatory signalling pathways. | 30 min.
  Musle and fat biopsies during a hyperinsulinaemic euglycaemic clamp (30 min. from the beginning of clamp)

CONTACTS AND LOCATIONS:
Overall Officials: Niels Møller, Professor, Principal Investigator — Aarhus University Hospital
Locations (1):
- Medical Department MEA, NBG, Aarhus University Hospital, Aarhus, Denmark

REFERENCES:
- [Derived] Bach E, Nielsen RR, Vendelbo MH, Moller AB, Jessen N, Buhl M, K-Hafstrom T, Holm L, Pedersen SB, Pilegaard H, Bienso RS, Jorgensen JO, Moller N. Direct effects of TNF-alpha on local fuel metabolism and cytokine levels in the placebo-controlled, bilaterally infused human leg: increased insulin sensitivity, increased net protein breakdown, and increased IL-6 release. Diabetes. 2013 Dec;62(12):4023-9. doi: 10.2337/db13-0138. Epub 2013 Jul 8. PMID 23835341